CLINICAL TRIAL: NCT06028412
Title: Comparison of Segmentectomy and Lobectomy in Small (2 Cm or Less 0.5<CTR<1) Non-small Cell Lung Cancer: a Prospective, Multicenter Randomized Controlled Study
Brief Title: Comparison of Sublobar and Lobectomy in Small (2 Cm or Less 0.5<CTR<1) Non-small Cell Lung Cancer: a Prospective, Multicenter Randomized Controlled Study
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Xiaolong Yan, Dr. (Other)
Responsible Party: Sponsor-Investigator, Xiaolong Yan, Dr., chief physician, Tang-Du Hospital
Organization: Tang-Du Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XKT-Y-20221121
Record Dates: First submitted 2023-08-29; First posted 2023-09-08 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: NSCLC, Stage I
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Anterior Temporal Lobectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sublobar (Experimental): The minimize unit is the subsegment, the subloar group includes wedge resection, subsegmentectomy, segmentectomy.
  It is recommended to perform intraoperative lymph node pathology (not mandatory). If lymph node metastasis is positive, we must switch to lobectomy+system lymph node dissection. lymph node sampling, selective lymph node dissection or systematic lymph node dissection are allowed in this group.
  Interventions: Procedure: Sublobar
- lobectomy (Placebo Comparator): lobectomy and Systematic lymph node dissection
  Interventions: Procedure: Lobectomy

INTERVENTIONS:
Procedure: Sublobar — The minimize unit is the subsegment, the subloar group includes wedge resection, subsegmentectomy, segmentectomy.
  It is recommended to perform intraoperative lymph node pathology (not mandatory). If lymph node metastasis is positive, we must switch to lobectomy+system lymph node dissection. lymph node sampling, selective lymph node dissection or systematic lymph node dissection are allowed in this group.
  Arms: Sublobar
Procedure: Lobectomy — lobectomy+system lymph node dissection
  Arms: lobectomy

SUMMARY:
The early NSCLC（Non-small cell lung cancer） patients with partial solid nodules mainly composed of solid components, whose maximum tumor diameter was ≤ 2.0cm and 0.5<CTR（Consolidation tumor ratio）<1, as indicated by preoperative thin slice CT, were selected as the study objects. The short-term and long-term effects of segmental resection and lobectomy under Thoracoscopy were compared to provide high-level evidence for the selection of surgical treatment methods for early NSCLC.

DETAILED DESCRIPTION:
Since Cahan reported on "radical lobectomy" in 1960, lobectomy has become the standard surgical method for lung cancer, and its efficacy has long been verified in clinical practice. In 2006, the National Comprehensive Cancer Network (NCCN) lung cancer diagnosis and treatment guidelines listed thoracoscopic lobectomy as one of the standard surgical methods for early non-small cell lung cancer (NSCLC) for the first time. However, in recent years, an increasing number of retrospective studies have found that the efficacy of subpulmonary lobectomy in treating stage IA NSCLC is similar to that of lobectomy. Not only is there no difference in survival rate, but perioperative complications and mortality are lower, and lung function is also more protected. Anatomical segmental lung resection was also recommended as one of the surgical options for early NSCLC patients by the US NCCN guidelines in 2010. With the development of thin-layer CT diagnosis and treatment technology, the detection rate of early lung cancer with main imaging manifestations such as small pulmonary nodules and ground glass nodules (GGO) has improved. The solid components in GGO are often considered as infiltrating components with a high possibility. The Lung Cancer Surgery Research Group (LCSSG) of the Japanese Clinical Oncology Group used Solid Component Ratio for ground glass nodules, which stratified the study population by the ratio of the maximum solid component diameter to the maximum tumor diameter, and began multiple clinical trials related to subpulmonary lobectomy, And these clinical trials will clarify whether subpulmonary lobectomy can be used as a standard surgical procedure for early NSCLC patients.

Among them, the recently released research results of the JCOG 0802 trial suggest that for peripheral NSCLC with tumor diameter ≤ 2cm and CTR>0.5, the segmental resection group even outperforms the lobectomy group in terms of 5-year OS as the main endpoint, which overturns people's understanding of early lung cancer surgery methods. The JCOG 0802 results showed that the local recurrence rate in the segmental resection group was 10.5%, while in the lobectomy group it was 5.4% (p=0.0018). However, the relatively high value of local recurrence in the segmental resection group did not result in a decrease in the final 5-year RFS and 5-year OS. And in the JCOG 0201 study, the tumor size of all recurrent cases within 5 and 10 years after surgery was ≥ 1cm, and the majority were patients with CTR=1.0. However, it is worth noting that the JCOG 0802 experiment also has corresponding problems: 1. The initial enrollment condition is CTR>0.25, and with the release of the long-term results of the JCOG 0201 experiment, the CTR value is adjusted from 0.25 to 0.5; 2. More than half of the enrolled patients have pure solid nodules (CTR=1.0); 3. During the research phase, preoperative 3D reconstruction technology was not used for surgical resection range planning. Therefore, the experimental results of JCOG 0802 deserve further in-depth research, and the choice of surgical methods for patients with partial solid nodules (PSN) with a diameter ≤ 2cm and a CTR<1 is also the most perplexing issue for thoracic surgeons at present. Someone has proposed that for PSN patients with a diameter ≤ 2cm, subpulmonary lobectomy surgery can replace traditional lobectomy surgery, and patients have similar prognosis. However, this theory is derived from retrospective studies and there is a lack of relevant prospective randomized controlled study data, which should be confirmed in prospective studies. Therefore, the issues raised in the above research pose key scientific questions for the implementation of this project: whether segmental resection of the lung has similar long-term survival and short-term efficacy to lobectomy for patients with partial solid nodules with a tumor diameter of ≤ 2cm and 0.5<CTR<1 requires a multicenter, prospective, non-inferiority, randomized controlled study to answer.

In summary, based on previous literature and clinical studies, this project conducted a multicenter, prospective, open, non-inferiority, randomized controlled study in conjunction with multiple well-known hospitals in China, targeting early NSCLC patients with partial solid nodules (different from JCOG 0802, excluding solid nodules with CTR=1) with a maximum tumor diameter of ≤ 2.0cm and a maximum tumor diameter of 0.5<CTR<1 on preoperative thin-layer CT. The main endpoint of the study was 5-year DFS, Compare the short-term and long-term efficacy of VATS pulmonary segment resection and lobectomy in the treatment of early NSCLC. The expected results of this project will further fill the gaps in previous clinical research and provide high-level evidence for the selection of surgical treatment methods for early NSCLC. It is expected to enrich or rewrite the current surgical treatment guidelines for lung cancer, improve the level of NSCLC surgical treatment, and have important theoretical significance and practical value.

ELIGIBILITY:
Inclusion Criteria:

* nitial inclusion criteria:

  1. Age 18-75 years old, regardless of gender;
  2. ECOG PS score 0-1 points (Attachment 3.4);
  3. Preoperative clinical staging for patients with suspected NSCLC lesions in Phase I (according to AJCC Eighth Edition staging standards, Attachment 3.5);
  4. Thin slice CT indicates that the maximum tumor diameter is ≤ 2.0cm;
  5. Pre operative CT prompts 0.5<CTR<1.0;
  6. Good lung function (FEV1>1.5 L or FEV1% ≥ 60%), able to tolerate both segmental resection and lobectomy;
  7. The number of pulmonary nodules that need to be processed is ≤ 3, and the nodules are located in the same side of the lung;
  8. Those who voluntarily sign the research informed consent form can comply with the research visit plan and other protocol requirements.

     Exclusion Criteria:

Initial exclusion criteria:

1. Hypertension and diabetes difficult to control;
2. Pregnant or lactating women;
3. Those who have received anti-tumor treatment (radiotherapy, chemotherapy, Targeted therapy, immunotherapy) before surgery;
4. Previous history of lung surgery;
5. Interstitial pneumonia, Pulmonary fibrosis or severe Emphysema;
6. Those who undergo thoracotomy or change the surgical plan due to various reasons during surgery;
7. Severe mental illness;
8. Individuals with a history of severe heart disease, heart failure, myocardial infarction, or angina within the past 6 months;
9. Active bacterial or fungal infections that are difficult to control;
10. Individuals who have conducted other clinical trials in the three months prior to enrollment.

Secondary exclusion criteria:

1. The postoperative pathological result was Benign tumor;
2. Postoperative pathological results of non NSCLC malignant tumors;
3. Non small cell lung cancer confirmed histologically during operation, but with malignant Pleural effusion and pleural dissemination

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 660 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
DFS(Disease-free survival) | Follow up for 5 years for all patients after enrollment
  Disease-free survival (DFS) is a number that tells the chances of staying free of a disease or cancer after a particular treatment. It is the percentage of individuals in the treatment group who are likely to be free of the signs and symptoms of a disease after a specified duration of time.

SECONDARY OUTCOMES:
OS (Overall survival) | Follow up for 5 years for all patients after enrollment
  The time between the onset of randomization and the occurrence (progression) or death (for any reason) of the tumor.
Pulmonary function test measure lung volume | Respectively measure lung function at the 6th and 12th months after surgery
  Pulmonary function test (PFTs) are noninvasive test that show how well the lungs are working after surgery.
Pulmonary function test measure rates of flow | Respectively measure lung function at the 6th and 12th months after surgery
  Pulmonary function test (PFTs) are noninvasive test that show how well the lungs are working after surgery.
Pulmonary function test measure gas exchange | Respectively measure lung function at the 6th and 12th months after surgery
  Pulmonary function test (PFTs) are noninvasive test that show how well the lungs are working after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: xiaolong yan, Principal Investigator — The Second Affiliated Hospital of Air Force Medical University University of PLA
Locations (1):
- The Second Affiliated Hospital of Air Force Medical University University of PLA, Xi'an, Shannxi, China

IPD SHARING:
Plan to Share IPD: Yes
The official website of the Second Affiliated Hospital of the Air Force Military Medical University of PLA（http://tdwww.fmmu.edu.cn/）
Supporting Information: Study Protocol
Time Frame: 2023 10years